CLINICAL TRIAL: NCT06072846
Title: An Alternative Approach to Fatigue and Comfort Levels in Hemodialysis Patients: Reiki Energy Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Merve Topac, Principal investigator, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NamikKU.
Record Dates: First submitted 2023-09-01; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Hemodialysis
Keywords: Chronic Renal Failure; Hemodialysis; Reiki; Therapy; Tiredness; Disease
MeSH Terms: conditions — Kidney Failure, Chronic; Fatigue; Disease

STUDY DESIGN:
Intervention Model Description: There is an initiative and control group. Reiki therapy will be provided to the intervention group. Monitoring will be performed on the control group.
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- enterprise group (Experimental): Reiki therapy will be applied to the initiative group. Evaluation will be carried out with pre-test and post-test
  Interventions: Behavioral: Reiki Energy Therapy
- Control group (No Intervention): The control group will not be interfered with. The control group will not be interfered with and will only be evaluated by pre-test and post-test by monitoring.

INTERVENTIONS:
Behavioral: Reiki Energy Therapy — Reiki Therapy will be applied to the intervention group
  Arms: enterprise group

SUMMARY:
Chronic renal failure (CRF) is a chronic and progressive kidney disease caused by impaired metabolic and endocrine functions as a result of a decrease in glomerular filtration rate (GFR), the role of the kidney in maintaining fluid electrolyte balance. KRG, which has high mortality and morbidity, is defined as an important public health problem due to the fact that it also causes a great burden on health systems.

Reiki is not an alternative to allopathic medicine; it is a "complementary" therapy that can be applied together with all other medical and therapeutic techniques. It has been reported that the deep relaxation created by Reiki relieves anxiety, stress and pain perception and promotes a feeling of psycho-spiritual well-being. Reiki strengthens the energy pathways and meridians, facilitates the natural process of healing. It regulates the energy systems of the body that are blocked by stress or a negative situation. Reiki, which is applied for various purposes, ensures that blood and lymph circulation continue in a healthy way, stimulates the autonomic nervous system. In this way, reiki facilitates physical and spiritual relaxation and strengthens health.

DETAILED DESCRIPTION:
Chronic renal failure (CRF) is a chronic and progressive kidney disease caused by impaired metabolic and endocrine functions as a result of a decrease in glomerular filtration rate (GFR), the role of the kidney in maintaining fluid electrolyte balance. KRG, which has high mortality and morbidity, is defined as an important public health problem due to the fact that it also causes a great burden on health systems.The development and stage of chronic kidney failure are related to the patient's symptoms and clinical signs. Patients are usually asymptomatic until stage 4-5. Symptoms of the disease generally begin with weakness. When the GFR falls below 30 ml/min, clinical signs are observed in the patient. No matter what stage of KRG is, dietary and pharmacological treatment methods are required. Renal replacement therapies are peritoneal dialysis, kidney transplantation and hemodialysis.

Hemodialysis treatment is the process of cleaning the blood taken from the patient by passing it into dialysis fluid through a semi-permeable membrane with the help of a machine to eliminate waste products that cannot be removed from the blood, such as creatinine, urea, in patients with end-stage renal failure, and returning it to the patient.

Difficulties and complications experienced in the adaptation process related to the disease and treatment in hemodialysis patients negatively affect patient comfort. Various methods have been used to reduce the symptoms experienced by hemodialysis patients and increase their comfort level. It has been found that complementary therapies such as aromatherapy, progressive relaxation exercises, music therapy, acupressure, massage therapy, reflexology, yoga and reiki, which hemodialysis patients use to relieve fatigue, have an effect on symptoms.

Difficulties and complications experienced in the adaptation process related to the disease and treatment in hemodialysis patients negatively affect patient comfort. Various methods have been used to reduce the symptoms experienced by hemodialysis patients and increase their comfort level. It has been found that complementary therapies such as aromatherapy, progressive relaxation exercises, music therapy, acupressure, massage therapy, reflexology, yoga and reiki, which hemodialysis patients use to relieve fatigue, have an effect on symptoms.

Reiki is not an alternative to allopathic medicine; it is a "complementary" therapy that can be applied together with all other medical and therapeutic techniques. It has been reported that the deep relaxation created by Reiki relieves anxiety, stress and pain perception and promotes a feeling of psycho-spiritual well-being.Reiki strengthens the energy pathways and meridians, facilitates the natural process of healing. It regulates the energy systems of the body that are blocked by stress or a negative situation. Reiki, which is applied for various purposes, ensures that blood and lymph circulation continue in a healthy way, stimulates the autonomic nervous system. In this way, reiki facilitates physical and spiritual relaxation and strengthens health.

ELIGIBILITY:
Inclusion Criteria:

1. Who is 18 years of age or older
2. Who has been receiving hemodialysis treatment for at least 6 months and receives 3.hemodialysis for at least 2 sessions per week

4.Without communication and mental problems 5.Who can speak Turkish 6.Who agrees to participate in the study

Exclusion Criteria:

1. Who is under the age of 18
2. Who has been receiving hemodialysis for less than 6 months
3. With communication and mental problems
4. Who cannot speak Turkish
5. Those who do not agree to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-09-04 (Estimated)

PRIMARY OUTCOMES:
Reiki Energy Therapy | 1 years
  The scales to be used are the Fatigue Severity Scale and Hemodialysis Comfort Scale II. With these scales Changes in fatigue and comfort levels will be expected in hemodialysis patients with reiki treatment.
  The Fatigue Severity Scale (YÖS): Krupp et al. it was developed by (1989) and the scale was developed by Armutlu et al. a Turkish validity and reliability study was conducted by Dec in 2003; Cronbach alpha value: 0.85 and consists of 9 items, each item is scored between 1-7 (1=I disagree at all, 7=I completely agree) and the total score is calculated by taking the average of 9 items. The average was determined as "<2.8; No fatigue, >6.1 ; I have Chronic Fatigue Syndrome". The lower the total score, the less fatigue.

SECONDARY OUTCOMES:
Hemodialysis Comfort Scale II (HKÖ) | 1 years
  Hemodialysis Comfort Scale II (HKÖ): This scale, developed by Coşar by conducting a literature review, is a 5-point likert type scale consisting of 26 items - six sub-dimensions. Substances that are not reversed on the scale (19, 20, 22, 25, 26) 1 from towards 5; inverse substances (1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 21, 23, 24) 5 it is scored from 1 to correct. Comfort increases as the scale score increases, comfort decreases as the score decreases. The items and December of points included in the sub-dimensions; Physical refreshment: 5, 6, 7, 8. (4-20 points) Physical relaxation: 1, 2, 3, 4. (4-20 points) Psychospirital relaxation: 18, 19, 20, 21, 22, 23, 24, 25, 26. (9-45 points) Psychospiritual empowerment: 14, 15, 16, 17. (4-20 points) Environmental empowerment: 12, 13. (2-10 points) Sociocultural relaxation: 9, 10, 11. (3-15 points) and the scale score December min - max= 26-130 points

CONTACTS AND LOCATIONS:
Overall Officials: Nurhan ÖZPANCAR ŞOLPAN, Principal Investigator — Namik Kemal University
Locations (1):
- Nurhan ÖZPANCAR ŞOLPAN, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang F, Liao M, Wang P, Liu Y. Cost-effectiveness analysis of renal replacement therapy strategies in Guangzhou city, southern China. BMJ Open. 2021 Feb 5;11(2):e039653. doi: 10.1136/bmjopen-2020-039653. PMID 33550227
- [Background] McManus DE. Reiki Is Better Than Placebo and Has Broad Potential as a Complementary Health Therapy. J Evid Based Complementary Altern Med. 2017 Oct;22(4):1051-1057. doi: 10.1177/2156587217728644. Epub 2017 Sep 5. PMID 28874060
- [Background] Bossi LM, Ott MJ, DeCristofaro S. Reiki as a clinical intervention in oncology nursing practice. Clin J Oncol Nurs. 2008 Jun;12(3):489-94. doi: 10.1188/08.CJON.489-494. PMID 18515247
- See also: The Current Status of Renal Replacement Therapies in Turkey: Turkish Society of Nephrology Registration Summary 2016 Report — https://turkjnephrol.org/en/current-status-of-renal-replacement-therapies-in-turkey-summary-of-turkish-society-of-nephrology-registry-2016-report-1627021
- See also: Comparing the Effects of Lavender Oil and Olive Oil Massage on Pain due to Muscular Cramp during Hemodialysis — https://bijps.uobaghdad.edu.iq/index.php/bijps/article/view/1235/927